CLINICAL TRIAL: NCT03810872
Title: An Open Explorative Phase II, Open Label Study of Afatinib in the Treatment of Advanced Cancer Carrying an EGFR, a HER2 or a HER3 Mutation
Brief Title: An Explorative Study of Afatinib in the Treatment of Advanced Cancer Carrying an EGFR, a HER2 or a HER3 Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AZ-VUB (Other)
Responsible Party: Principal Investigator, Dr. Lore Decoster, Coordinator Investigator, AZ-VUB
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Precision 2 - 1200.264
Record Dates: First submitted 2019-01-12; First posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Cancers Harbouring an EGFR Mutation, (Excluding Non-squamous Non- Small Cell Lung Cancer, a Registered Indication), a HER2 Mutation or a HER3 Mutation
MeSH Terms: interventions — Afatinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open label (Other): Afatinib 40 mg/day during Period 1 Afatinib 40 mg/day + Paclitaxel 80mg/kg/3w during Period 2
  Interventions: Drug: Afatinib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Afatinib — Open label
Drug: Paclitaxel — Paclitaxel

SUMMARY:
Objective(s):To investigate the efficacy and safety of afatinib in EGFR, HER 2 and HER3 mutated cancers, regardless of cancer type, excluding EGFR mutated non-small cell lung cancer.

Methodology:Open label, genomic driven trial (basket trial)

No. of patients total entered:Optimal Simon two stage design for the three genetic driven cohorts: 10 patients will be enrolled per cancer type in the first stage and an additional 19 in the second stage (maximum total 87 patients)

Indication : cancers harbouring an EGFR mutation(excluding non-squamous non- small cell lung cancer, a registered indication), a HER2 mutation or a HER3 mutation

Test product(s) : Afatinib At progression paclitaxel will be added for those patients that have no contra-indications

dose: Starting dose of afatinib at 40 mg/day. Dose increase to 50 mg in the absence of adverse events. Stepwise dose reduction to 30,20, 10 mg/day according to drug-related adverse events.

At progression, addition of paclitaxel 80 mg/m2 weekly 3w/4 to afatinib 40 mg/day .

mode of admin. : Oral for afatinib Intravenous for paclitaxel

Duration of treatment: Continuous treatment until progression or unacceptable adverse events or withdrawal of consent.

At disease progression, add paclitaxel until progression or unacceptable adverse event or withdrawal of consent if no contra-indications.

Criteria for efficacy: Primary Endpoint:

• Response rate (CR+ PR) via RECIST v1.1

Secondary Endpoints:

* Disease control rate (CR+PR+SD)
* Progression free survival
* Overall survival
* To correlate tumor response with findings on tumor biopsies
* To investigate resistance mechanisms
* response rate (CR+ PR) determined by RECIST and progression free survival on the combination therapy of afatinib and paclitaxel

Criteria for safety: Incidence and intensity of adverse events according CTCAE v4.0

ELIGIBILITY:
Inclusion Criteria:

* Women and men with locally advanced or metastatic cancers harboring either an activating EGFR mutation or a HER2 mutation or a HER3 mutation
* Failure of at least one line of standard systemic therapy
* No eligibility for other open genomic driven phase I, II or III trial available for these tumor genotypes
* ECOG performance status ≤2
* Patient with a life expectancy >3 months
* Patients able to provide written informed consent prior to enrollment into the clinical trial.
* Adequate organ function

Exclusion Criteria:

* Non squamous non-small cell lung cancer harbouring an EGFR mutation (registered indication)
* Chemotherapy, biological therapy or investigational agents within four weeks prior to the start of study treatment
* Known hypersensitivity to afatinib or the excipients of any of the trial drugs
* Prior treatment with afatinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2017-06-21 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | 6 weeks
Incidence and intensity of adverse events | 4 weeks

SECONDARY OUTCOMES:
Disease control rate | 6 weeks
Progression free survival | 6 weeks
Overall survival | 6 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- Belgium (5):
  - Institut Jules Bordet, Brussels
  - Les Cliniques Universitaires St Luc, Brussels
  - Universitaire Ziekenhuis Antwerpen, Edegem
  - UZ Gent, Ghent
  - CHU Sart-Tilman, Liège

IPD SHARING:
Plan to Share IPD: No